CLINICAL TRIAL: NCT05968911
Title: Survival and Predictive Factors of Clinical Outcome in Patients With Acquired Brain Injury
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Michal Soták, Principal Investigator, Charles University, Czech Republic
Other Study IDs: ABI_UVN
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Acquired Brain Injury
Keywords: acquired brain injury; consciousness disorders; prognosis; persistent vegetative state
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma brain injury: Patients with acquired brain injury of traumatic etiology.
- Non-trauma brain injury: Patients with acquired brain injury of non-traumatic etiology.

SUMMARY:
The prediction of the final neurological and functional status of patients with acquired brain injury remains very uncertain despite the findings of current medicine. The aim of the study is to evaluate the clinical outcomes in patients with the most severe degree of brain injury hospitalized in the long-term intensive care unit of the Military University Hospital Prague.

DETAILED DESCRIPTION:
The prediction of the final neurological and functional status of patients with acquired brain injury remains very uncertain despite the findings of current medicine. Current medical knowledge is particularly limited in patients with the most severe brain injury who had to be tracheostomized and admitted to long-term intensive care unit. In the Czech Republic, there is a complete lack of data on clinical outcomes in these patients.

Some recent studies has not confirmed the long-standing better outcome in patients with traumatic brain injury compared to non-traumatic etiologies. The aim of the study is to evaluate the clinical outcomes in patients with the most severe degree of brain injury hospitalized in the long-term intensive care unit of the Military University Hospital Prague.

ELIGIBILITY:
Inclusion Criteria:

* Acquired brain injury
* Initial Glasgow Coma Scale (GCS) score less than 8 points
* Tracheostomy for persistent impairment of consciousness

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the long-term intensive care unit of the University Hospital Prague in years 2015-2022 with acquired brain injury of the five most common etiologies (traumatic injury, ischemic stroke, intracerebral hemorrhage, subarachnoid haemorrhage, anoxic injury), whose initial Glasgow Coma Scale was less than 8 points and were tracheostomized due to persistent impairment of consciousness.
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Level of consciousness achieved | three months
  Initial Glasgow coma scale (GCS) and GCS at discharge. Minimal points 3, maximal point 15. The higher the score the better the outcome.
Level of self-sufficiency | three months
  Initial level of self-sufficiency and self-sufficiency at discharge using Barthel score.
  0-100 points. A patient scoring 100 points is continent, feeds himself, dresses himself, gets up out of bed and chairs, bathes himself, walks at least a block, and can ascend and descend stairs.
  A score of 0 means that the patient does not meet any of the activities described above.

SECONDARY OUTCOMES:
Length of survival after discharge from intensive care. | three months
  Length of survival after discharge from intensive care. In days.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Trtíková, Mgr., Ph.D., Study Chair — CHARLES UNIVERSITY, FIRST FACULTY OF MEDICINE AND GENERAL UNIVERSITY HOSPITAL IN PRAGUE
Locations (1):
- Military University Hospital Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wabl R, Williamson CA, Pandey AS, Rajajee V. Long-term and delayed functional recovery in patients with severe cerebrovascular and traumatic brain injury requiring tracheostomy. J Neurosurg. 2018 Jul 6;131(1):114-121. doi: 10.3171/2018.2.JNS173247. Print 2019 Jul 1. PMID 29979120
- [Background] Magliacano A, De Bellis F, Panico F, Sagliano L, Trojano L, Sandroni C, Estraneo A. Long-term clinical evolution of patients with prolonged disorders of consciousness due to severe anoxic brain injury: A meta-analytic study. Eur J Neurol. 2023 Dec;30(12):3913-3927. doi: 10.1111/ene.15899. Epub 2023 Jun 8. PMID 37246500
- [Background] Multi-Society Task Force on PVS. Medical aspects of the persistent vegetative state (1). N Engl J Med. 1994 May 26;330(21):1499-508. doi: 10.1056/NEJM199405263302107. PMID 7818633